CLINICAL TRIAL: NCT06214637
Title: Effectiveness of Melissa Officinalis in Various Concentrations for the Treatment of Probable Sleep Bruxism in Children and Adolescents: Controlled and Randomized Clinical Trial
Brief Title: Effectiveness of Melissa Officinalis for the Treatment of Probable Sleep Bruxism in Children and Adolescents
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Larissa Soares Lima da Silva, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 69209423.4.0000.0268
Record Dates: First submitted 2023-12-12; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Sleep Bruxism; Adolescent; Children; Temporomandibular Joint Disorders
Keywords: Sleep bruxism; Homeopathy; Adolescent; Children
MeSH Terms: conditions — Sleep Bruxism; Temporomandibular Joint Disorders | interventions — lemon balm leaf extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): It will be administered for a period of 30 days, once a day before bed, with a 15-day wash-out interval. The placebo, a drug without active substance, that will be administered to research participants will be the biotherapeutic vehicle, that is, 30% alcohol (v/v), which is commonly used as a vehicle for homeopathic medicines.
  Interventions: Drug: Placebo
- Melissa officinalis 6 CH (Experimental): It will be administered for a period of 30 days, once a day before bed, with a 15-day wash-out interval. This concentration that will be administered to research participants will be the biotherapeutic vehicle, that is, 30% alcohol (v/v), which is commonly used as a vehicle for homeopathic medicines.
  Interventions: Drug: Melissa
- Melissa officinalis 9 CH (Experimental): It will be administered for a period of 30 days, once a day before bed, with a 15-day wash-out interval. This concentration that will be administered to research participants will be the biotherapeutic vehicle, that is, 30% alcohol (v/v), which is commonly used as a vehicle for homeopathic medicines.
  Interventions: Drug: Melissa
- Melissa officinalis 12 CH (Experimental): It will be administered for a period of 30 days, once a day before bed, with a 15-day wash-out interval. This concentration that will be administered to research participants will be the biotherapeutic vehicle, that is, 30% alcohol (v/v), which is commonly used as a vehicle for homeopathic medicines.
  Interventions: Drug: Melissa

INTERVENTIONS:
Drug: Melissa — The test solutions will be administered once a day through administration in drops for children between 5 and 10 years old and for adolescents between 11 and 16 years old. As participants will be between 5 and 16 years old, children will be given a minimum of 5 and a maximum of 10 drops of the solutions per individual (Tavares-Silva, Holandino et al. 2019) as well as a maximum of 10 drops for adolescents of solutions per individual (Taylor, Lancaster et al. 2000). Highlighting that the prescription of Melissa officinalis will be at night, around 20/30 minutes before bedtime, respecting the indications for the medications described in the Hahnemannian Materia Medica (Vijnovsky, 2003). All medications must be taken away from meals and they will be instructed not to use mentholated substances, respecting a minimum time of 30 minutes.
  Arms: Melissa officinalis 12 CH; Melissa officinalis 6 CH; Melissa officinalis 9 CH
Drug: Placebo — It will be administered for a period of 30 days, once a day before bed, with a 15-day wash-out interval. The placebo, a drug without active substance, that will be administered to research participants will be the biotherapeutic vehicle, that is, 30% alcohol (v/v), which is commonly used as a vehicle for homeopathic medicines.
  Arms: Placebo

SUMMARY:
Objective: To investigate, through a controlled and randomized clinical trial, the effectiveness of using Melissa officinalis in different concentrations in the treatment of children and adolescents with probable sleep bruxism. Methodology: This is a randomized, triple-blind, crossover, and placebo-controlled clinical trial. The research participants will be children aged 5 to 10 years old and adolescents aged 11 to 16 years old who attend dental treatment at the FO/UFRJ Pediatric Dentistry Clinics. After approval by the Human Research Ethics Committee, children and adolescents will undergo homeopathic treatment with Melissa officinalis in different concentrations for possible sleep bruxism. In addition, research participants will undergo an assessment of TMJ, sleep, circadian cycle, quality of life, and quality of life related to oral health. The data will be tabulated and analyzed according to sex, age group, presence of possible sleep bruxism, presence or absence of TMD, circadian characteristics, presence or absence of sleep disorders, daytime and nighttime behavioral characteristics. The data will be tabulated and evaluated using SPSS 21.0. Absolute and relative frequency, odds ratio, correlation analysis and other relevant analyzes and statistical tests (p<0.05) will be carried out in accordance with the objectives proposed by the study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 to 16 years;
* Patients with complete primary dentition, mixed or secondary dentition;
* Patients with probable sleep bruxism.

Exclusion Criteria:

* Patients with special needs (psychological, psychiatric and neurological, diagnosed with anxiety disorder or any systemic impairment);
* Patients with parafunctional habits (finger sucking and/or pacifier, onychophagia, biting objects, etc.)
* Patients with caries lesions in dentin in one or more elements (ICDAS values 4, 5 and 6);
* Patients affected by molar-incisor hypomineralization (MIH)
* Patients with dental anomalies such as dentinogenesis imperfecta, amelogenesis imperfecta, dysplasia dentin, hypoplasia, and enamel hypocalcification;
* Patients with severe malocclusions: Class II and III or crossbite and open bite type;
* Patients using orthodontic appliances;
* Patients who are taking medications for anxiety disorders or any other that cause alterations in the central nervous system or that alter salivary flow.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
General objective | Twice a month
  Number of participants who had a positive response to the proposed treatment, that is a reduction in bruxism episodes during the sleep period.

CONTACTS AND LOCATIONS:
Overall Officials: Lucianne Cople Maia, Phd, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The results will be released after the completion of the clinical trial, which forms part of the responsible researcher's Phd thesis.